CLINICAL TRIAL: NCT04975061
Title: A Phase 2 Clinical Study of YY-20394 in Patients With Relapsed/Refractory Thymic
Brief Title: A Phase 2 Clinical Study of YY-20394 in Patients With Relapsed/Refractory Thymic Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: YY-20394-011
Record Dates: First submitted 2021-07-12; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Effectiveness，Safety，Thymic Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: YY-20394 — YY-20394 is a small molecule inhibitor.

SUMMARY:
This study is a single-arm, open, multi-center phase II clinical trial, the main purpose of which is to evaluate the effectiveness and safety of YY-20394 in the treatment of patients with relapsed/refractory thymic cancer.

The research adopts the Simon two-stage design method, which is carried out in two stages.

DETAILED DESCRIPTION:
This study is a single-arm, open, multi-center phase II clinical trial, the main purpose of which is to evaluate the effectiveness and safety of YY-20394 in the treatment of patients with relapsed/refractory thymic cancer.

The research adopts the Simon two-stage design method, which is carried out in two stages.

The first stage:

In the first phase, a single-arm, open, multi-center study was adopted, and YY-20394 monotherapy was given to patients who met the enrollment conditions. The trial enrolled 18 subjects. If ≥2 subjects had ORR (clinical benefit), then enter the second phase, otherwise the trial will be terminated.

The second stage:

Refer to the efficacy data of the first phase to decide whether to conduct the second phase of clinical research.

In the second phase, a single-arm, open, multi-center study was adopted. Patients who met the enrollment conditions were given YY-20394 monotherapy. In the second phase, 40 subjects will continue to be enrolled.

A total of 58 subjects were included in the two stages. During the study period, the investigator judged the best curative effect of all subjects according to the response evaluation criteria in solid tumours (Response evaluation criteria in solid tumours, RECIST 1.1). IRC will use the same standards to evaluate the efficacy of the imaging results of all subjects, and the entire review process will be conducted in accordance with an independent review procedure. The Research Safety Monitoring Committee (SMC) will continue to review the safety of study drugs. SMC will be responsible for monitoring safety data and making decisions on research-related issues, such as study enrollment, dose selection, whether to continue the study, etc.

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18 years old and above;
2. Patients with thymic cancer confirmed histologically (WHO classification), including all subtypes;
3. Inoperable advanced disease (Masaoka-Koga staging), which progresses after receiving at least one systemic chemotherapy;
4. Volunteer to participate in this clinical trial, understand the research procedures and be able to sign written informed consent;
5. ECOG performance status (PS) level 0 to 1;
6. Estimated survival time ≥ 3 months;
7. According to the RECIST1.1 standard, the patient has at least one measurable lesion;
8. Be able to provide tissues from archive tissue samples or newly obtained core or excision biopsy tissues of tumor lesions;
9. According to the judgment of the investigator, it can comply with the test plan;
10. Past anti-tumor therapy (including chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy) from the end to the first use of the study drug washout period ≥ 4 weeks, including oral fluorouracil and small molecule targeted drugs Washout period ≥ 2 weeks;
11. Good organ function level:

    1. Bone marrow function needs to meet:

       * Absolute neutrophil count (ANC) ≥1.5×109/L;
       * Platelet count (PLT) ≥80×109/L;
       * Hemoglobin (Hb) ≥9 g/dL;
    2. Liver function

       * Serum total bilirubin (TBIL) ≤1.5 x ULN (except for Gilbert syndrome, total bilirubin ≤2.5 x ULN);
       * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0×ULN (or recorded liver transfer: 5.0×ULN);
    3. Kidney function

       • Serum creatinine clearance rate (CrCl) ≤1.5 x ULN OR ≥60ml/min (calculated according to Cockcroft-Gault formula);
    4. Coagulation function

       • International normalized ratio (INR) ≤ 1.5 × ULN, unless the subject is receiving anticoagulant therapy, as long as the PT or PTT is within the expected therapeutic range of the anticoagulant; activated partial thrombin time (APTT) ≤ 1.5 × ULN, Unless the subject receives anticoagulant therapy, as long as the PT or PTT is within the expected therapeutic range of the anticoagulant;
    5. Heart function • Ejection fraction (LVEF) ≥50%; Fridericia method corrected QT interval (QTcF) male <450ms, female <470ms.

Exclusion Criteria:

1. Suffer from thymic cancer that can be cured by surgery or radiation;
2. Those who have used anti-tumor drugs targeting PI3Kδ have progressed (such as being out of the group due to intolerance) outer);
3. Suffer from ongoing malignant tumors or other malignant tumors that require active treatment. Skin base Bottom cell carcinoma, except for squamous cell carcinoma of the skin or cervical cancer in situ after potential treatment;
4. Known active central nervous system (CNS) metastasis/cancerous meningitis. Previously accepted Subjects of brain metastasis therapy can participate as long as they are stable (there is no evidence of imaging progress at least 4 weeks before the first dose of trial treatment, and any neurological symptoms have returned to baseline levels), and there are no new or enlarged Evidence of brain metastases in patients, and have not used steroids for at least 7 days before the trial treatment;
5. Suffered from active autoimmune disease in the past 3 months and required systemic treatment, or Documented history of clinically severe autoimmune disease, or syndrome requiring systemic steroids or immunosuppressive agents. Except subjects with vitiligo or childhood asthma/atherosclerosis, subjects who need intermittent bronchodilators or topical steroid injections, and subjects with hypothyroidism and stable to hormone replacement or Sjorgen syndrome;
6. Those who have active viral, bacterial or fungal infections and need treatment (such as pneumonia, etc.);
7. According to the judgment of the investigator, there is a serious harm to the safety of the patient, or affect the completion of the research The accompanying diseases of the study (such as uncontrollable hypertension, uncontrollable diabetes, active interstitial lung disease, etc.);
8. People with allergies, or those who are known to have a history of allergies to the components of this medicine;
9. The baseline pregnancy test of pregnant women, lactating women, or women with childbearing potential is positive;
10. Have a history of immunodeficiency, including HIV test positive, or have other acquired, congenital Sexual immunodeficiency disease, or history of organ transplantation, or allogeneic bone marrow or hematopoietic stem History of cell transplantation;
11. Previously suffering from heart diseases, including: (1) angina pectoris; (2) those requiring clinical intervention Arrhythmia; (3) Myocardial infarction; (4) Heart failure; (5) Other researched Other heart diseases judged to be unsuitable for participating in this trial;
12. Skin basal cell carcinoma and uterine cancer that have been cured of other malignant tumors in the past 5 years Except for cervical carcinoma in situ;
13. People with HBV or HCV infection (defined as HbsAg and/or HbcAb positive and HBV DNA copy number ≥1×104 copy number/ml or ≥2000 IU/ml) or acute or chronic active hepatitis C (HCV) antibodies Positive;
14. Live vaccine has been vaccinated within 30 days before the first dose of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically confirmed thymic cancer (WHO classification), including all subtypes; inoperable advanced disease (Masaoka-Koga staging); progressed after receiving at least one systemic chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 6 months
  Overall response rate consists of complete response and partial response